CLINICAL TRIAL: NCT01087710
Title: Effect of Novel Medical Food on Reducing the Frequency and Severity of Asthma Symptoms and Airway Hyper-responsiveness in Children With Mild to Moderate Persistent Asthma
Brief Title: Effect of Medical Food on Reducing Asthma Symptoms in Asthmatic Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Bobbie Swearengin, Director, Abbott Nutrition
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK22
Record Dates: First submitted 2010-03-08; First posted 2010-03-16 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2010-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — gamma-carboxyglutamyl-gamma-carboxyglutamic acid; Vitamins; Minerals

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- novel nutritional formula (Experimental)
  Interventions: Other: medical food with EPA and GLA, vitamins and minerals
- Control nutritional product (Active Comparator): 1 8oz serving per day for 12 weeks
  Interventions: Other: medical food minus EPA and GLA, antioxidant vitamins/minerals

INTERVENTIONS:
Other: medical food with EPA and GLA, vitamins and minerals — 1 8oz serving per day for 12 weeks
  Arms: novel nutritional formula
Other: medical food minus EPA and GLA, antioxidant vitamins/minerals — 1 8oz serving a day for 12 weeks
  Arms: Control nutritional product

SUMMARY:
To determine the effect of medical food on reducing asthma symptoms in asthmatic children.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children who have had mild to moderate persistent asthma for at least 1 year and are between 6 and 14 years of age, and not currently being treated with steroids are eligible.

Each subject also has to have:

* Subject is off of controller therapy 4 wks preceding visit 1.
* Mild to moderate persistent asthma
* Methacholine responsiveness with an FEV1 PC20
* Able to perform reproducible spirometry
* Verbal assent in addition to consent
* History of prior clinical varicella or varicella vaccine.
* Nonsmoker in past year.

Exclusion Criteria:

* Asthma symptoms and/or albuterol use consistent with severe persistent asthma during the run-in period.
* Subject with FEV1 < 80% predicted at visit 1 or FEV1 < 70% predicted at visit 2.
* Two or more hospitalizations for asthma in the past year.
* Subject has received oral, nasal, inhaled, or IM corticosteroids during the preceding month.
* Subject has received leukotriene modifiers, theophylline derivatives, or mast cell stabilizers for asthma within 4 weeks before visit 1
* Subject is receiving one or more of the following medications:

  * Astemizole prior to 3 months of visit 1
  * Oral, inhaled or parenteral corticosteroids prior to 4 weeks of visit 1
  * Cromolyn, antimuscarinics, cimetidine, metoclopramide, phenobarbital, phenytion, terfenadine, loratadine, or anticholingeric agents prior to 2 weeks of visit 1.
  * Theophylline prior to 4 weeks of visit 1
* Subject with active upper respiratory tract infection prior to 4 weeks before visit 1
* Subject with acute sinus disease requiring antibiotic treatment within 1 week before visit
* Subject with an emergency department treatment for asthma within 1 month, prior intubation for asthma, or hospitalization for asthma within 3 months
* Subject has known bleeding disorder and/or is on medication known to have significant anticoagulant effects.
* Subject has known hypersensitivity to any of the ingredients
* Subject is taking either pill, powder, or liquid forms of nutritional and/or health food supplements within the past 4 weeks prior to visit
* Subject unable to tolerate or unwilling to take the full dose of the nutritional study formulas
* Cystic fibrosis or any other chronic lung disease other than asthma.
* Subject having gastroesophogeal reflux undergoing medical treatment
* Significant medical illness other than asthma that could require oral corticosteroids during the study.
* Subject is receiving allergen hyposensitization therapy other than an established maintenance regimen
* Subject has received IV globulins or immunosuppressants.
* Subject is known to be human immunodeficiency virus (HIV) positive.
* Pregnancy or lactation.
* If of child bearing potential, failure to practice abstinence or use of an acceptable birth control method.
* Subject is morbidly obese

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2004-07; Primary Completion 2005-12 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
asthma free days | 12 weeks

SECONDARY OUTCOMES:
reduction of airway hyper-responsiveness | 12 weeks
time to the first asthma exacerbation | 12 weeks
respiratory function (spirometry) | 12 weeks
need for rescue for exacerbations of asthma symptoms. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stehen DeMichele, PhD, Study Chair — Abbott Nutrition
Locations (1):
- National Jewish Health, Denver, Colorado, United States

REFERENCES:
- [Derived] Covar R, Gleason M, Macomber B, Stewart L, Szefler P, Engelhardt K, Murphy J, Liu A, Wood S, DeMichele S, Gelfand EW, Szefler SJ. Impact of a novel nutritional formula on asthma control and biomarkers of allergic airway inflammation in children. Clin Exp Allergy. 2010 Aug;40(8):1163-74. doi: 10.1111/j.1365-2222.2010.03523.x. Epub 2010 Jun 7. PMID 20545703